CLINICAL TRIAL: NCT02274909
Title: PILATES AND PNF METHODS INDUCES SIMILAR STRENGTH GAINS, BUT DIFFERENT NEUROMUSCULAR ADAPTATIONS IN ELDERLY WOMEN
Brief Title: Pilates and PNF Methods Induces Similar Strength Gains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do PiauÍ (Other)
Responsible Party: Principal Investigator, FABIANA TEIXEIRA DE CARVALHO, UESPI, Universidade Estadual do PiauÍ
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UESPI-8
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Sarcopenia
Keywords: electromyography; aged; muscle strength; wavelet analysis; pilates; proprioceptive neuromuscular facilitation
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention): The subjects received no intervention and continued with their daily activities.
- Pilates group (Active Comparator): The exercise protocol of Pilates method consisted of muscle stretching of the upper limbs, trunk and lower limbs before the exercises. Then, exercises involving range of motion and strength of upper limbs, trunk and lower limbs were performed, always associated with breathing in different positions and with increasing repetitions and resistance along the weeks of training.
  Interventions: Other: TRAINING PROGRAM
- PNF group (Active Comparator): The exercises from the PNF method were performed with stretching, associated to hold-relax technique, for upper and lower limbs. Then, subjects carried out exercises with the upper limbs, in a bilaterally symmetrical pattern, and with the lower limbs, in the asymmetric bilateral pattern. Additionally, scapular and pelvic girdle exercises were done with symmetrical and reciprocal combination.
  Interventions: Other: TRAINING PROGRAM

INTERVENTIONS:
Other: TRAINING PROGRAM — Sixty healthy elderly women were randomly divided into 3 groups: Pilates group (PG), PNF group (PNFG) and Control group (CG). Pilates and PNF groups underwent one-month training program with Pilates and PNF methods, respectively. CG received no intervention along the one month.
  Arms: PNF group; Pilates group

SUMMARY:
To compare the influence of a training program with Pilates and PNF methods to elderly women on the strength gains and motor control during voluntary contractions

DETAILED DESCRIPTION:
Sixty healthy elderly women were randomly divided into 3 groups: Pilates group (PG), PNF group (PNFG) and Control group (CG). Pilates and PNF groups underwent one-month (three times per week) training program with Pilates and PNF methods, respectively. CG received no intervention along the one month. The maximal isometric force from knee extension and flexion, as well as the EMG signal from quadriceps and biceps femoris were recorded before and after the one-month intervention period. A two-way analysis of variance (3 groups x 2 measures) was used to compare the results from EMG signal, isometric force and force variability and force spectrum. A one-month training program with Pilates and PNF methods induces similar strength gains from knee flexors and extensors, without differences between methods, but PG exhibited greater low gamma drive (i.e., 30-60 Hz band) after the training period. Both Pilates and PNF methods were efficient to improve the muscle strength, but with different neuromuscular adaptations in elderly women. These results give support to the recommendation these methods to older age groups, since the increment of lower limb muscle strength is important for gait, postural stability and performance of daily life activities of this population.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects were between 60 an 80 years old, sedentary and healthy

Exclusion Criteria:

* Subjects were excluded from the study if they presented any orthopedic, neurological, cardiac, vestibular, visual, or psychiatric impairment which would not allow them to perform all the tasks in the study

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
EMG measurement | WERE MEASUREMENT BEFORE AND ONE MONTH, IN ALL PARTICPANTS